CLINICAL TRIAL: NCT05447702
Title: A Single-arm, Prospective Phase II Study of Camrelizumab Plus Apatinib and Chemotherapy as Neoadjuvant Therapy for Triple Negative Breast Cancer (TNBC)
Brief Title: Study of Camrelizumab Plus Apatinib and Chemotherapy as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shuangyue Liu, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-026
Record Dates: First submitted 2022-06-30; First posted 2022-07-07 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; apatinib; 130-nm albumin-bound paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Apatinib + Chemotherapy (Experimental): Participants received neoadjuvant therapy with four 4-week cycles of camrelizumab (200 mg, q2w) plus apatinib (250 mg, qd) and nab-paclitaxel (125 mg/m2, qw), followed by four 2-week cycles of camrelizumab (200 mg, q2w) plus apatinib (250 mg, qd) and epirubicin (90 mg/m2, q2w) + cyclophosphamide (600 mg/m2, q2w).
  Interventions: Drug: Camrelizumab; Drug: Apatinib; Drug: Nab-paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Camrelizumab — Intravenous (IV) infusion
Drug: Apatinib — po.
Drug: Nab-paclitaxel — IV infusion.
Drug: Epirubicin — IV infusion.
Drug: Cyclophosphamide — IV infusion.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of camrelizumab in combination with apatinib and chemotherapy as neoadjuvant therapy in participants with triple negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer.
* 18-75 Years, female.
* Early or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression).
* Tumor stage: II-III.
* ECOG Performance Status of 0-1.
* life expectancy is not less than 3 months.
* at least one measurable lesion according to RECIST 1.1.
* Adequate hematologic and organ function.
* Must be willing to use an adequate method of contraception for the course of the study.

Exclusion Criteria:

* Stage Ⅳ (metastatic) breast cancer or bilateral breast cancer.
* Inflammatory breast cancer.
* Has received prior any anti-tumor therapy within the past 12 months prior to signing informed consent, including chemotherapy, targeted therapy, radiation therapy, immunotherapy, biotherapy and TAE.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], and/or anti-VEGFR agent.
* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Major surgical procedure within 4 weeks prior to initiation of study treatment.
* Has a history of autoimmune disease.
* Has a history of hypertension that not well controlled by antihypertensive treatment
* Has a history of myocardial infarction, severe/unstable angina pectoris, NYHA Class 2 or above cardiac insufficiency, clinically significant supraventricular or ventricular arrhythmia, or symptomatic congestive heart failure within the last 6 months.
* Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases.
* Administration of a live attenuated vaccine within 28 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B, Hepatitis C or Autoimmune hepatitis.
* Severe infections within 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment.
* Has evidence of active tuberculosis within 1 year prior to initiation of study treatment.
* Prior allogeneic stem cell or solid organ transplantation.
* Peripheral neuropathy grade ≥2.
* Has clinically significant intestinal obstruction.
* Arterial/venous thrombosis events that occurred within 3 months before enrollment, such as cerebrovascular accidents, deep vein thrombosis, or pulmonary embolism.
* Has hemoptysis symptoms within 2 months before enrollment and the maximum daily hemoptysis ≥ 2.5 ml.
* Clinically significant bleeding symptoms or clear bleeding tendency occurred within 3 months before enrollment.
* Has known genetic or acquired bleeding or thrombotic tendency.
* Abnormal coagulation (INR>1.5 or APTT>1.5 x ULN) with bleeding tendency, receiving thrombolysis or anticoagulation therapy, or requiring long-term antiplatelet therapy.
* Has a known hypersensitivity to the components of the study treatment or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial.
* History of neurological or psychiatric disorders, including epilepsy or dementia.
* Any other situation evaluated by researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pCR rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 28 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive tumor on hematoxylin and eosin evaluation of breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.

SECONDARY OUTCOMES:
pCR rate using the definition of ypT0/Tis (i.e., absence of invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement) at the time of definitive surgery | Up to approximately 28 weeks
  pCR rate (ypT0/Tis) is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants.
Objective Response Rate (ORR) | Up to approximately 28 weeks
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until definitive surgery or disease progression.
Event-Free Survival (EFS) | Up to approximately 3 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Invasive Disease-Free Survival (iDFS) | Up to approximately 3 years
  iDFS events are defined as follows: (1) Ipsilateral invasive breast tumor recurrence. (2) Ipsilateral local-regional invasive breast cancer recurrence. (3) Ipsilateral second primary invasive breast cancer. (4) Contralateral invasive breast cancer. (5) Distant recurrence. (6) Death attributable to any cause.
Adverse events (AEs) | Up to approximately 37 weeks
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Luo, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China